CLINICAL TRIAL: NCT03243383
Title: A Pilot Trial to Prevent Hospital Readmission of Patients With Diabetes
Brief Title: Readmission Prevention Pilot Trial in Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24306; 5K23DK102963 (NIH)
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
Keywords: readmission
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-risk Group (No Intervention): Low-risk as determined by the predicted risk of readmission by the DERRI. The low-risk group will be followed in a prospective, observational arm of the study.
- High-risk Group - Intervention (Experimental): High-risk as determined by the predicted risk of readmission by the DERRI. Subjects in the high-risk group will be randomly assigned to receive either the intervention (DiaTOHC Program) or usual care (control).
  Interventions: Other: DiaTOHC Program
- High-risk Group - Usual Care (No Intervention): Patients in the high-risk usual care group will receive the standard hospital discharge process and post-discharge followup.

INTERVENTIONS:
Other: DiaTOHC Program — 1. Patient-centered education 1a) Standardized diabetes discharge instructions and education 1b) Comprehensive discharge plan review
  2. Peri-discharge coordination of care
  3. A1c-based adjustment of diabetes therapy
  4. Post-discharge support
  Arms: High-risk Group - Intervention

SUMMARY:
Post-discharge hospital utilization, i.e., readmissions within 30 days of discharge (30d readmissions) and emergency department (ED) visits, are a high-priority quality measure and target for cost reduction. Patients with diabetes are disproportionately over-represented in 30d readmissions, especially among racial minorities and urban populations. We have developed and validated a tool, the Diabetes Early Readmission Risk Indicator (DERRI), to predict 30d readmission risk among diabetes patients, which is a critical prerequisite for targeting limited resources for reducing readmission risk to those most in need. Currently, there are no proven interventions to reduce the risk of 30d readmission specifically among patients with diabetes. This proposal will assess the feasibility and acceptability of a novel, multifactorial intervention, the Diabetes Transition of Hospital Care Program (DiaTOHC), designed to reduce post-discharge hospital utilization rates in a pilot randomized controlled trial. The intervention will include inpatient diabetes and discharge education, comprehensive discharge planning and coordination of care, A1c-based adjustment of diabetes therapy, and post-discharge support. Hospitalized patients with diabetes identified as high risk for readmission based on the DERRI will be randomized to the intervention or the control group, which will receive usual care. Such work is highly relevant in the current era of soaring health care costs and national health care reform.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes, defined by pre-admission use of a diabetes-specific medication and/or documentation of the diagnosis in the medical record.

Exclusion Criteria:

1. Age < 18 years at the time of admission
2. Female subjects who are pregnant and/or admitted to an obstetric service
3. Current or expected admission to a critical care unit
4. Binge drinking (5 or more alcoholic drinks for males or 4 or more alcoholic drinks for females on the same day) or drug abuse within 3 months before admission
5. Inpatient death
6. Transfer to another hospital or subacute facility
7. Discharge to hospice or a long-term care facility
8. Discharge expected within 12 hours or admission to a short-stay unit
9. Lack of access to a phone
10. Living more than 30 miles away from Temple University Hospital (TUH)
11. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of initial hospital readmission | Within 30 days after discharge
  The number of initial hospital readmissions will be recorded.

SECONDARY OUTCOMES:
Time to first readmission | Assessed at 30 days of discharge
  The time to first readmission will be recorded.
Incidence of emergency department (ED) visits | Assessed at 30 days of discharge
  The number of ED visits will be recorded.
A composite of 30 day readmission and ED visits | Assessed at 30 days of discharge
  The composite of 30 day readmission and ED visits will be calculated and recorded.
Incidence of primary care and specialist provider follow-up visits scheduled and attended | Assessed at 30 days of discharge
  The number of primary care provider follow-up visits scheduled and attended will be recorded.
Incidence of medication review or reconciliation post-discharge | Assessed at 30 days of discharge
  The number of medication reviews or reconciliations post-discharge will be recorded.
Cost of post-discharge care as a sum of ED visits, readmission, and PCP visits | Assessed at 30 days of discharge
  The cost of post-discharge care as a sum of ED visits, readmission, home health services, and outpatient provider visits
Cost of the intervention | Assessed at 30 days of discharge
  The cost of nurse and physician time.
Subject experience assessed by a brief questionnaire | Assessed at 30 days of discharge
  Subject experience via a brief questionnaire will be assessed.
Self-monitored blood glucose levels and frequency of testing | Assessed at 30 days of discharge
  Number of blood glucose tests per day and incidence of hypoglycemia.
Change in well-being | Baseline to 5 weeks after discharge
  Change in well-being from baseline to 5 weeks after discharge as measured by the World Health Organization Well-Being Index (WHO-5)
Change in diabetes-related distress | Baseline to 5 weeks after discharge
  Change in diabetes-related distress at 5 weeks after discharge as measured by the Problem Areas in Diabetes (PAID) scale
Change in perceived social support | Baseline to 5 weeks after discharge
  Change in perceived social support at 5 weeks after discharge as measured by the Multidimensional Scale of Perceived Social Support (MSPSS)
Change in perceived stress | Baseline to 5 weeks after discharge
  Change in perceived stress at 5 weeks after discharge as measured by the perceived stress scale (PSS)
Change in diabetes knowledge | Baseline to 5 weeks after discharge
  Change in diabetes knowledge at 5 weeks after discharge as measured by the Diabetes Knowledge Test (DKT2)
Change in A1c level | Baseline to 3 months discharge
  The change in A1c level from baseline to 3 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rubin, MD, MSc, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubin DJ, Handorf EA, Golden SH, Nelson DB, McDonnell ME, Zhao H. DEVELOPMENT AND VALIDATION OF A NOVEL TOOL TO PREDICT HOSPITAL READMISSION RISK AMONG PATIENTS WITH DIABETES. Endocr Pract. 2016 Oct;22(10):1204-1215. doi: 10.4158/E161391.OR. PMID 27732098
- [Background] Rubin DJ. Hospital readmission of patients with diabetes. Curr Diab Rep. 2015 Apr;15(4):17. doi: 10.1007/s11892-015-0584-7. PMID 25712258
- [Background] Rubin DJ, Donnell-Jackson K, Jhingan R, Golden SH, Paranjape A. Early readmission among patients with diabetes: a qualitative assessment of contributing factors. J Diabetes Complications. 2014 Nov-Dec;28(6):869-73. doi: 10.1016/j.jdiacomp.2014.06.013. Epub 2014 Jun 28. PMID 25087192
- See also: Diabetes Early Readmission Risk Indicator (DERRI) — https://redcap.templehealth.org/redcap/surveys/?s=3XCPCAMKWE

DOCUMENTS (2):
  • Study Protocol (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT03243383/Prot_001.pdf
  • Informed Consent Form (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT03243383/ICF_002.pdf